CLINICAL TRIAL: NCT05168618
Title: AtezoCab: A Phase II Study of Cabozantinib in Combination With Atezolizumab in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC) With Non-Measurable Disease
Brief Title: Cabozantinib and Atezolizumab for the Treatment of Metastatic Castration-Resistant Prostate Cancer, The AtezoCab Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI143814; NCI-2021-13110 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI143814 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — atezolizumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cabozantinib, atezolizumab) (Experimental): Patients receive cabozantinib PO QD on days 1-21 and atezolizumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Cabozantinib S-malate

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184

SUMMARY:
This phase II trial tests whether cabozantinib and atezolizumab work to shrink tumors in patients with castrate-resistant prostate cancer that had spread to other places in the body (metastatic). Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cabozantinib and atezolizumab may kill more tumor cells in patients with metastatic castrate-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the disease control rate in metastatic castration-resistant prostate cancer (mCRPC) patients with non-measurable disease as assessed by Prostate Cancer Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the combination as measured by prostate-specific antigen (PSA) progression-free survival (PFS).

II. To evaluate the efficacy of the combination as measured by PSA 50% response rate.

III. To evaluate the efficacy of the combination as measured by radiographic progression-free survival (PFS).

IV. To evaluate the efficacy of the combination as measured by overall survival (OS).

V. To evaluate the safety of cabozantinib S-malate (cabozantinib) in combination with atezolizumab in patients with mCRPC with non-measurable disease.

EXPLORATORY OBJECTIVE:

I. To analyze tissue and tumor-based biomarkers to evaluate the mechanisms of treatment activity and resistance.

OUTLINE:

Patients receive cabozantinib orally (PO) once daily (QD) on days 1-21 and atezolizumab intravenously (IV) over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months until disease progression or start of another therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male subject aged >= 18 years
* Histologically or cytologically confirmed prostatic adenocarcinoma without small cell histology
* Metastatic disease progression after continuous androgen deprivation therapy for hormone sensitive state
* Patient must have non-measurable disease outside the pelvis (above aortic bifurcation) per RECIST 1.1 criteria. Non-measurable disease can be bone lesions and/or extraskeletal disease
* Disease progression on or after at least one prior novel hormonal therapy (NHT) (defined as second-generation antiandrogen therapies that include but are not limited to abiraterone acetate, enzalutamide, apalutamide, darolutamide)
* Eastern Cooperative Oncology Group (ECOG) performance Status =< 2
* Effective castration with serum testosterone levels =< 0.5 ng/mL (=<1.7 nmol/L)
* Tumor tissue available (archival or recent tumor biopsy). If no tumor tissue is available, patients can be enrolled after approval from Principal Investigator.
* Absolute neutrophil count (ANC) >= 1500/mm^3 without granulocyte colony-stimulating factor support
* White blood cell count >= 2500/uL
* Lymphocyte count >= 0.5 x 10^9/L (500/uL)
* Platelet count >= 100,000/mm^3 without transfusion in the 2 weeks prior to cycle 1 day 1 (C1D1)
* Hemoglobin >= 9 g/dL
* Serum albumin >= 2.5 g/dl
* For patients not receiving therapeutic anticoagulation: prothrombin time (PT)/International normalized ratio (INR) or partial thromboplastin time (PTT) test < 1.5 x institutional upper limit of normal (ULN). For patients receiving therapeutic anticoagulation: stable anticoagulant regimen as determined by Investigator
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN). For subjects with Gilbert's disease =< 3 x institutional ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional ULN

  * Subjects with liver metastases will be allowed to enroll with AST and ALT levels =< 5 x institutional ULN
* Alkaline phosphatase (ALP) =< 3 × institutional ULN. Patients with documented liver or bone metastases: ALP =< 5 x institutional ULN
* Serum creatinine =< 1.5 x institutional ULN or calculated creatinine clearance >= 40 mL/min by Cockcroft-Gault formula
* Urine protein/creatinine ration (UPCR) =< 1mg/mg (=< 113.2 mg/mmol), or 24-hour (h) urine protein =< 1 g
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 5 months after the last dose of study treatment
* Male subjects must agree to use a condom during intercourse for the duration of study therapy
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) v5.0 from toxicities related to any prior cancer therapy, unless considered clinically not significant by the treating investigator and/or stable on supportive therapy
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines
* Capable of understanding and complying with the protocol requirements

Exclusion Criteria:

* Prior chemotherapy in the metastatic castration refractory prostate cancer setting is not allowed (taxane-based in metastatic castration-sensitive disease is allowed)
* Prior treatment with cabozantinib, CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-a, anti-PD1 and anti-PD-L1 therapeutic antibodies
* Prior treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment
* Receiving other investigational agents
* Patients with measurable disease outside the pelvis (above aortic bifurcation) per RECIST 1.1 criteria
* History of Leptomeningeal disease
* Uncontrolled tumor-related pain

  * Note: Patients requiring pain medication must be on a stable regimen at study entry
  * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Major surgery (e.g., laparoscopic nephrectomy, gastrointestinal (GI) surgery, removal or biopsy of brain metastasis) within 4 weeks before first dose of study treatment or anticipation of need for a major surgical procedure during the study. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival [OS] rate > 90%), such as locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast
* Known brain metastases or cranial epidural disease

  * Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before the first dose of study treatment after radiotherapy or at least 4 weeks prior to the first dose of study treatment after major surgery (e.g. removal or biopsy of brain metastasis) will be allowed on trial. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the first dose of study treatment
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines), low-dose low molecular weight heparins (LMWH), or prophylactic dose of anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban.
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Administration of a live, attenuated vaccine (e.g., FluMist) within 30 days before first dose of any study treatment and for 5 months after the last dose of any study treatment
* Current evidence of uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class II, III or IV, unstable angina pectoris, serious unstable cardiac arrhythmias
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), other ischemic events, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before the first dose of study treatment

      * Subjects with a diagnosis of incidental, sub segmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation for at least 1 week before first dose of study treatment
    * Uncontrolled hypertension defined as persistent systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg despite optimal antihypertensive treatment
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
* Lesions invading or encasing any major blood vessels
* Any active or history of known or suspected autoimmune disease as determined to be clinically significant by treating investigator's clinical judgement will be excluded , including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis (see Appendix for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

  * Controlled Type 1 diabetes mellitus who are an insulin regimen
  * Autoimmune-related hypothyroidism who are on thyroid replacement hormone
  * Skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
  * Conditions not expected to recur in the absence of an external trigger
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before first dose of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
  * Note: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Any active infection requiring systemic treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) or oral valacyclovir (valaciclovir) are eligible for the study
* Acute or chronic hepatitis B or C infection, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection. Note: Subjects on effective HIV antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Serious non-healing wound/ulcer/bone fracture
* Malabsorption syndrome
* Uncompensated/symptomatic hypothyroidism
* Moderate to severe hepatic impairment (Child-Pugh B or C)
* Requirement for hemodialysis or peritoneal dialysis
* History of solid organ or allogenic stem cell transplant
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

  * Note: Patients with indwelling catheters (e.g., PleurX) are allowed
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | At 24 weeks
  Measured per Prostate Cancer Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 with a 95% confidence interval.

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA) progression-free survival (PFS) | From treatment initiation until documented clinical or radiographic progression or death from any cause, assessed up to 3 years
  Kaplan-Meier methods will be used to analyze PFS and will be presented with 95% confidence intervals. PSA progression is defined by PCWG3 criteria.
PSA levels | Baseline up to 30 days after completion of study treatment
  Will be monitored per treatment schedule to assess the proportion of patients with a 50% reduction in PSA levels (PSA50) compared to the baseline value at the time of study enrollment.
Progression-free survival (PFS) | From the start date of treatment and the date of first recurrence or death from any cause, assessed up to 3 years after the initiation of therapy
  Kaplan-Meier methods will be used to analyze PFS and will be presented with 95% confidence intervals. Measured with RESIST 1.1.
Overall survival | From trial initiation and death of any cause, assessed up to 5 years
  Will be evaluated for survival using Kaplan-Meier estimation.
Incidence of adverse events (AEs) | Up to 30 days after completion of study treatment
  The severity of the AEs will be graded according to the Common Terminology Criteria for Adverse Events version 5.0. The statistical analysis of the safety data will be descriptive and tabular.

CONTACTS AND LOCATIONS:
Overall Officials: Umang Swami, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No